CLINICAL TRIAL: NCT06357897
Title: Faculty of Medicine, Chulalongkorn University
Brief Title: The Efficacy and Palatability of Developed Polyethylene Glycol-based Formula for Children With Functional Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Duc Long Tran, Principal investigator of Center of Excellence in Clinical Virology, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0093/67
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Functional Constipation
Keywords: Functional constipation; Children; Polyethylene glycol; Palatability

STUDY DESIGN:
Intervention Model Description: Intervention group received PEG-Chula Control group received Forlax
Who Masked: Participant, Care Provider, Investigator
Masking Description: The intervention and control were prepared in the similar sachet and was blinded to investigatiors, participants and guardians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEG-Chula (Experimental): PEG-Chula is developed from local PEG 4000 used at King Chulalongkorn Memorial Hospital (KCMH) with the addition of sweetener and flavours and prepared into sachets labelled A, B, C and D.
  Interventions: Drug: Local PEG4000
- Standard PEG (Other): Standard PEG (Forlax) is prepared into the sachets labelled A, B, C and D with similar packaging and appearance.
  Interventions: Drug: Commercial PEG4000

INTERVENTIONS:
Drug: Local PEG4000 — PEG-Chula is developed from PEG 4000 used at King Chulalongkorn Memorial Hospital with added sweetener and flavours. Children will be given PEG-Chula at a dose of 0.5 - 1 g/kg/day.
  Other Names: PEG-Chula
  Arms: PEG-Chula
Drug: Commercial PEG4000 — For commercial PEG, We use Forlax as the control group. Children will be given Forlax at a dose of 0.5 - 1 g/kg/day.
  Other Names: Forlax
  Arms: Standard PEG

SUMMARY:
This study aims to evaluate the efficacy and palatability of a developed polyethylene glycol-based formula compared with the standard polyethylene glycol (PEG) in the treatment of children with functional constipation for 8 weeks. Besides, we also aim to assess the side effects of a developed PEG-based formula as well as evaluate the change of rectal diameter from baseline at each visit between 2 groups.

DETAILED DESCRIPTION:
Total 52 children age 6 months to 18 years old diagnosed with functional constipation will be enrolled in this study. They will be randomised in Group A or Group B.

Children in group A will receive PEG-Chula at a dose of 0.5 - 1 g/kg/day for a duration of 56 days.

Children in group B will receive the standard PEG formula (Forlax) at a dose of 0.5 - 1 g/kg/day for a duration of 56 days.

PEG-Chula and standard PEG will be prepared in sachets with similar packaging and appearance labelled A, B, C, D.

Children in both groups will also receive counseling on toilet training, water intake, and fiber intake in the same manner.

Parents will be advised to record symptoms, dietary intake, and dose of medication in a logbook.

Children will visit the researchers on days 7, 14, 28, and 56 to collect data on symptoms, stool diameter, bowel size measured by ultrasound, side effects, and medication compliance. Children with poor compliance will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

Children will be enrolled in this study when they meet 2 criteria:

* Age from 6 months to 18 years old
* Children are diagnosed with FC according to ROME IV criteria

Exclusion Criteria:

Children will be excluded from the study if they meet any of the following criteria:

* Having an organic cause of constipation such as anorectal malformations, Hirschsprung disease, myelomeningocele, hypothyroidism, etc.
* Suspected GI obstruction
* Receiving medication affecting bowel movement
* Having a history of allergy to PEG and stevia.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The frequency of stool | At 7 days, 14 days, 28 days and 56 days
  The frequency of stool per day
Stool consistency assessed by Bristol stool chart | At 7 days, 14 days, 28 days and 56 days
  The Bristol stool chart has 7 pictures of stool appearance. The number 1 mean hard stool and number 7 mean watery stool

SECONDARY OUTCOMES:
Fecal incontinence | At 7 days, 14 days, 28 days and 56 days
  Number of fecal incontinence occurs per day
Rectal diameter | At 7 days, 14 days, 28 days and 56 days
  The rectal diameter was measured by abdominal USG
Adverse events | At 7 days, 14 days, 28 days and 56 days
  Adverse events (i.e diarrhea, abdominal pain, bloating, nausea or vomiting)
Palatability of medication assessed by facial Hedonic scale | At 7 days, 14 days, 28 days and 56 days
  The facial Hedonic scale contains 5 pictures of facial expression and number 1 mean dislike very much while number 5 means like very much

CONTACTS AND LOCATIONS:
Overall Officials: Palittiya Sintusek, Ph.D., Study Chair — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The data were collected anonymous.